CLINICAL TRIAL: NCT04388761
Title: Feasibility and Safety of Allogeneic Adipose Mesenchymal Stem Cells (aMSCs) Delivery Into Kidney Allografts Procured From Deceased Donors With High Kidney Donor Profile Index (KDPI)
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Challenges in recruiting participants.
Sponsor: Tambi Jarmi (Other)
Responsible Party: Sponsor-Investigator, Tambi Jarmi, Principal Investigator, Mayo Clinic
Organization: Mayo Clinic (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20-000264
Record Dates: First submitted 2020-05-12; First posted 2020-05-14 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Ischemia Reperfusion Injury
MeSH Terms: conditions — Reperfusion Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Intra parenchymal injection (Experimental): 5 subjects will receive AMSCs via direct injection into the kidney parenchyma only
  Interventions: Drug: Allogeneic adipose derived mesenchymal stem cells
- Intra-arterial infusion (Experimental): 5 subjects will receive AMSCs via intra-arterial infusion only
  Interventions: Drug: Allogeneic adipose derived mesenchymal stem cells
- Intra parenchymal injection & Intra-arterial infusion (Experimental): 5 subjects will receive AMSCs via direct injection into the kidney parenchyma and intra-arterial infusion
  Interventions: Drug: Allogeneic adipose derived mesenchymal stem cells

INTERVENTIONS:
Drug: Allogeneic adipose derived mesenchymal stem cells — Injection of Allogeneic adipose derived mesenchymal stem cells into the Kidney allograft

SUMMARY:
The purpose of this research is to test an investigational drug called Adipose Mesenchymal Stem Cells (aMSCs) for the treatment of ischemia re-perfusion injury (IRI) in patients that have had a kidney transplant.

ELIGIBILITY:
Inclusion Criteria:

* Male or female kidney transplant candidates age 18 and above.
* Patient is receiving kidney allograft from deceased donor with KDPI>85%.
* Ability of subject to give appropriate consent.
* Females of childbearing potential with agreement to use birth control for six months post-transplant.
* Approved by the Mayo Clinic Transplant Selection Committee.
* Signed Authorization for Donation of Anatomical Gifts on file.

Exclusion Criteria:

* Positive pregnancy test at the time of the kidney offer is called for the potential recipient.
* Kidney transplant potential recipients with active malignancy (except none melanoma skin malignancies).
* Patients with previous history of solid organ transplant (Heart, Lung, Intestine, Kidney and/or Pancreas).
* Patients with previous history of bone marrow transplant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-09 (Estimated); Primary Completion 2024-02 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
Serious Adverse Events (SAEs) | 1 year
  Number of serious adverse events reported. SAEs will include delayed graft function (30 days post-transplant), difficult to control bleeding (intraoperative), sub-scapular kidney hematoma or arteriovenous fistula formation (24 hours postop), and development of stroke, myocardial infarction, or pulmonary embolism (1 year post-transplant).

CONTACTS AND LOCATIONS:
Overall Officials: Tambi Jarmi, MD, Principal Investigator — Mayo Clinic

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials